CLINICAL TRIAL: NCT03698851
Title: Assessment of the Accuracy of the Clinical Parameters and Radiographs in Determining the Topography of Implant Bony Lesions
Brief Title: Assessment of the Accuracy of the Clinical Parameters & Radiographs in Determining the Topography of Implant Bony Lesions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to the difficulty in identifying suitable participants.
Sponsor: National Dental Centre, Singapore (Other)
Collaborators: Sunstar, Inc. (Industry)
Responsible Party: Principal Investigator, Tan Wah Ching, Dr, Visiting Specialist (Peridontics), Department of Restorative Dentistry, National Dental Centre, Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 253/2017
Record Dates: First submitted 2018-08-21; First posted 2018-10-09 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Peri-Implantitis
Keywords: Peri-Implantitis lesion; Dental Implants
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Guidor® and Guidor easy-graft® CRYSTAL Regeneration of the lesion will be performed with a synthetic membrane (Guidor®) with either Guidor easy-graft® CRYSTAL (Test).
  Interventions: Device: Guidor® and Guidor easy-graft® CRYSTAL
- Control Group (C) (Active Comparator): Guidor® and Guidor easy-graft® CLASSIC Regeneration of the lesion will be performed with a synthetic membrane (Guidor®) with either Guidor easy-graft® CLASSIC (Test).
  Interventions: Device: Guidor® and Guidor easy-graft® CLASSIC

INTERVENTIONS:
Device: Guidor® and Guidor easy-graft® CRYSTAL — A compound of biphasic calcium phosphate, 60 % hydroxyapatite and 40 % beta-tricalcium phosphate. The beta-tricalcium phosphate component completely resorbs via physiological dissolution in 5-15 months, while the interconnected hydroxyapatite remains embedded in the implantation site and forms an integrated long term osteoconductive scaffold with new bone.
  Arms: Test Group
Device: Guidor® and Guidor easy-graft® CLASSIC — Phase-pure beta-tricalcium phosphate that offers complete resorption via physiological dissolution in 5-15 months. This material has been used in oral surgery for more than 25 years and there are extensive research available on it.
  Arms: Control Group (C)

SUMMARY:
In recent years, dental implants have gained popularity as the treatment choice for replacement of missing teeth. With this, one of the late biological complications that arise is peri-implantitis. Based on a consensus conference in 2008, peri-implantitis was found in 28% and ≥ 56% of subjects and in 12% and 43% of implant sites (Zitzmann & Berglundh 2008). Detection of peri-implantitis is currently based on clinical parameters like probing depths and radiographic findings of bone loss. There is however no study that assess the variability of clinical probing and radiographic reading in relation to the true outline of the peri-implantitis lesion. The present study will measure variability of clinical probing and radiographs in relation to the true outline of the peri-implantitis lesion, as well as assess the use of 2 different bone substitutes in regenerating the lesions with a barrier membrane.

DETAILED DESCRIPTION:
Identification of peri-implant bony lesions by clinical parameters or radiographs alone may sufficiently reflect the topographical outline of a peri-implant bony lesion. To date, no comparative studies are available that identify the accuracy of clinical parameters or radiographs in outlining the extent and the severity of the lesion. If these parameters are of sufficient accuracy, surgical procedures to regenerate the lesion may be more predictable to plan.

The study population will be patients undergoing regular implant maintenance care in the National Dental Centre Singapore, Periodontics Unit, Department of Restorative Dentistry and yielding peri-implantitis (residual probing depths ≥6mm and bleeding on probing, bone loss of ≥2mm documented on periapical radiographs).

In the first part of the study, the variability of the clinical parameters and periapical radiographs will be assessed and compared to the actual bony lesions revealed after surgical access. This prospective cohort study will encompass 24 subjects. In the second part of the study, a randomised controlled clinical trial will be staged exploring the clinical outcomes of regenerative therapy of the peri-implant lesions applying 2 different bone substitutes with a barrier membrane for the principle of guided bone regeneration (GBR).

First part of study:

The null hypothesis is that of no difference in the mesial and distal radiographic readings as compared to the measurement obtained by clinical probing of the actual peri-implant lesions. The null hypothesis is also that of no difference between probing depth measurements and the actual lesions measured under open access.

Second part of study:

The null hypothesis is that of no difference in clinical outcomes with the use of a synthetic membrane (Guidor®) with a compound of biphasic calcium phosphate, 60 % hydroxyapatite and 40 % beta-tricalcium phosphate (Guidor easy-graft® CRYSTAL) (test) when compared to the same membrane and phase-pure beta-tricalcium phosphate (Guidor easy-graft® CLASSIC ) (control), in GBR of peri- implantitis lesions.

End Points - Efficacy For the subjects, the potential benefits may include improvement in the clinical outcomes.

End Points - Safety The risks involved include complications that may result with all surgeries, i.e., risk of infection, swelling, pain and bruising.

ELIGIBILITY:
Inclusion Criteria:

1. Medically healthy adults (ASA classification I-II), at least 21 years of age.
2. Diagnosed with peri-implantitis (at least one site with PPD of ≥ 6 mm, a positive bleeding on probing (BOP) and radiographic bone loss of ≥ 2 mm).
3. Had non-surgical therapy performed previously
4. Ability to comply with 6-month study follow-up.

Exclusion Criteria:

1. Medically compromised subjects (ASA classification III-V).
2. Had not gone through non-surgical therapy
3. Known allergy or other severe adverse reactions to the synthetic membrane and bone substitutes.
4. Self declared pregnancy or intend to conceive.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
The accuracy of clinical probing pocket depths to the true outline in peri-implantitis lesions | 6 months after GBR
  To determine the accuracy of clinical probing pocket depths (in mm) to the true outline in peri-implantitis lesions
The accuracy of peri-apical radiographic readings to the true outline in peri-implantitis lesions | 6 months after GBR
  To determine the accuracy of peri-apical radiographic readings (in mm) to the true outline in peri-implantitis lesions
Absolute change from baseline of probing pocket depth (PPD in mm) and the degree of bone fill at re-entry (6 months) | 6 months after GBR
  - To determine:
  1. Absolute change from baseline of probing pocket depth (PPD in mm) 6 months following GBR therapy in test and control
  2. The degree of bone fill at re-entry (6 months), as well as radiographically (in mm) following GBR

CONTACTS AND LOCATIONS:
Overall Officials: WAH CHING TAN, Principal Investigator — National Dental Centre, Singapore
Locations (1):
- National Dental Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided